CLINICAL TRIAL: NCT00854243
Title: Therapy Monitoring in Early Rheumatoid Arthritis: The Role of Greyscale and Power Doppler Sonography A Prospective Study Of 20 Egyptian Rheumatoid Arthritis Patients
Brief Title: Role of Greyscale and Power Doppler Sonography in Therapy Monitoring in Early Rheumatoid Arthritis (RA)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Ghada El-Mardenly, Cairo University
Other Study IDs: RA1
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the role of musculoskeletal ultrasound and power Doppler in early therapy monitoring of rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults: age at disease onset >18 years and < 50 years
* Disease duration < 3 month
* Fulfilling ARA criteria for classification of RA
* DMARD naive

Exclusion Criteria:

* Age at diagnosis < 18 years
* Disease duration > 3 month
* Previous use of DMARDS
* Previous use of biologics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult onset Rheumatoia Arthritis patients with a disease duration of less than 3 months
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)